CLINICAL TRIAL: NCT04986228
Title: DigiPuR: Digitally Supported Psychotherapy and Reintegration of Children and Adolescents With Mental Disorders After Inpatient Psychiatric Treatment
Brief Title: DigiPuR: Digitally Supported Psychotherapy and Reintegration
Acronym: DigiPuR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Universität Tübingen (Other)
Responsible Party: Principal Investigator, PD Dr. Annette Conzelmann, Head of the research department of the Department of Child and Adolescent Psychiatry, Psychosomatics and Psychotherapy at the University Hospital Tuebingen, University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 53-5400.1-005/09
Record Dates: First submitted 2021-05-28; First posted 2021-08-02 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Mental Disorder in Childhood
Keywords: Aftercare; E-Mental Health; Mental disorders; Triad; Adolescent; Child; Discharge; Readmission; Relapse prevention; Ambulatory assessment; Patient reported outcomes
MeSH Terms: conditions — Neurodevelopmental Disorders; Mental Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of two groups. One group will be offered regular follow-up consultations in the clinic (Control group). The other group will receive a digital aftercare service, consisting of video calls and an app, for a period of up to eight weeks after discharge (Intervention group). These enable an uncomplicated and yet intensive exchange with the clinic from the comfort of the participants' own homes. To enable to optimally plan the treatment and assess its success, all participants complete questionnaires on multiple time points about different topics.
Who Masked: Outcomes Assessor
Masking Description: Masking is only possible for data analysis, but not for participants, therapists, and study staff, because treatment is different in the two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital aftercare (Experimental): The group with the new digital aftercare is compared with the active control group with regular aftercare.
  Interventions: Other: Digital aftercare
- Treatment-as-usual (TAU) (Active Comparator): The group with regular aftercare (TAU) serves as an active control group.
  Interventions: Other: TAU

INTERVENTIONS:
Other: Digital aftercare — The intervention group will receive a digital aftercare service, consisting of video calls and an app, for a period of up to eight weeks after discharge. These enable an uncomplicated and yet intensive exchange with the clinic from the comfort of the participants' own homes. To enable to optimally plan the treatment and assess its success, all participants complete questionnaires on multiple time points about different topics.
  Arms: Digital aftercare
Other: TAU — The control group will receive the regular follow-up consultations in the clinic (treatment-as-usual, TAU). This includes at least one consultation with the case-leading therapist from the previous inpatient stay about 6 weeks after discharge. The assessment consisting of questionnaires at multiple time points about different topics is the same as in the intervention group.
  Arms: Treatment-as-usual (TAU)

SUMMARY:
The study "DigiPuR" (Digitally Supported Psychotherapy and Reintegration) examines the effectiveness of a new, digital aftercare program for children and adolescents after a psychiatric hospitalization in the intervention group compared to regular aftercare in the control group. Thereby, the randomized controlled trial with a naturalistic parallel group study design provides longitudinal data on the reintegration phase with a pre-post follow-up assessment and a daily ambulatory assessment from the point of view of patients, parents, and teachers. The aim of the new aftercare program is to facilitate reintegration after an inpatient hospital stay for children and adolescents as well as their attachment figures, to reduce readmissions and, if necessary, to ensure a good transition to outpatient structures. For this purpose, regular video calls without travel time between the children and adolescents as well as their attachment figures such as parents and teachers and, if necessary, external support systems are conducted with the clinic. Beyond these appointments, a smartphone-based secure messenger will allow all participants to communicate directly with the therapist. It is expected that the aftercare program in the intervention group will lead to improvements in health-related quality of life and treatment satisfaction, as well as reduce symptom severity and readmissions.

DETAILED DESCRIPTION:
Sample: All children and adolescents who were treated as partial or full inpatients in the Department of Child and Adolescent Psychiatry, Psychosomatics and Psychotherapy at the University Hospital Tuebingen, Germany as well as a primary attachment figure (parent or caregiver from a residential group) can participate in the study. Optionally, one or more teachers from the child's or adolescent's home school may also participate. The aim is to include N = 50 triplets (total sample about 150 persons) with 50 children and adolescents (n = 25 per group) and one attachment figure and one teacher each. The sample size was based on current RCT studies in this field as well as on the discharge numbers of the department.

Interventions: Participants will be assigned to one of two groups after informed written consent using a randomization list.

Intervention group: In the intervention group, 6 no longer than 50-minute video calls take place between the family and the case-leading therapist of the previous inpatient treatment (weekly until 4 weeks after discharge, then biweekly until 8 weeks after discharge). In order to adapt the aftercare to the needs of the patients, the case-leading therapist decides on the duration of the sessions as well as their participants (patients and/or parents and/or external support systems). The case-specific different contents are linked to the previous inpatient, behavioral therapy-oriented treatment with focus on the transfer of learned strategies into daily life. If patients and parents have agreed to the participation of teachers, three separate 30-45-minute video or telephone conferences are additionally conducted with one or more teachers from the home school and the case-leading therapist in the period up to 8 weeks after discharge. In addition, a handbook with the titel "Mental Illness in the School Environment" was developed, which enables teachers further information and support. Beyond the sessions with the case-leading therapists, the children and adolescents, parents and teachers have the opportunity to clarify content-related questions or organizational matters with the therapist via a secure messenger system on their own smartphone. Emergencies, on the other hand, are handled via the emergency number of the responsible clinic.

Control group: In the control group, the regular aftercare (treatment-as-usual) of the Department takes place. The regular aftercare usually includes a 50-minute follow-up consultation with the case-leading therapist in the clinic about 6 weeks after discharge.

Assessments: The assessments are the same in both groups.

Pre-Post-FollowUp: The admission and discharge assessment as part of the standard hospital assessment will be conducted using paper questionnaires (where necessary in exceptional cases online) by trained staff during the inpatient hospital stay in the period from preliminary talk on admission to one week after admission and in the period from one week before discharge to discharge (pre). For the post, follow-up 1, and follow-up 2 assessments (8, 24, and 37 weeks after discharge), participants receive an email with a link to an online survey that they can complete at home for one week using the browser on their computer, tablet, or smartphone. At each assessment point, the survey takes no longer than about 45 minutes to complete.

Ambulatory Assessment: The ambulatory assessment consists of questions about well-being, relationships, and the school situation that are answered daily from two weeks before to eight weeks after discharge in approximately 5 minutes between 5 and 9 in the evening by the children and adolescents, the participating attachment figure, and, if teachers participate, a teacher from the home school on their own smartphone. Teachers answer the questions only on school days and are given a larger time frame to respond to increase compliance. The questions for children and adolescents are presented in written and audiovisual form allowing children who are not yet confident readers to have the questions read aloud. Children and adolescents, parents, and teachers are reminded of daily questioning through alerts and can postpone alerts three times. Data collected in the ambulatory assessment is analyzed individually on a weekly basis by summarizing and graphing all responses. This overview of the patient's answers during the previous week(s) can be used by the case-leading therapist as a basis for the next regular video call.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents who received partial or full inpatient treatment in the Department of Child and Adolescent Psychiatry, Psychosomatics and Psychotherapy at the University Hospital Tuebingen, Germany (diagnosis irrelevant) and a relevant primary attachment figure (parent or caregiver from a residential group)
* Optionally teachers from the child's or adolescent's home school
* Participation in the study by a caregiver from a residential group and/or teachers from the home school always requires the written consent of the child or adolescent and his or her legal guardians
* Sufficient German language skills

Exclusion Criteria:

* Children and adolescents or the attending attachment figure who do not speak or understand the German language
* In case of acute psychological strain during the course of the study, an emergency presentation will take place at the responsible hospital. In case of an inpatient stay of less than two weeks, the study participation is continued, in case of more than two weeks, discontinued.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 61 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Change in symptom severity (patient report) | Admission, Pre (at discharge), Post (8 weeks after discharge), FollowUp1 (24 weeks after discharge), FollowUp2 (37 weeks after discharge)
  Symptom severity as assessed by patients is measured using the Diagnostic System for Mental Disorders according to ICD-10 and DSM-5 for Children and Adolescents - III Screening questionnaire (DISYPS-III SCREEN; Döpfner & Görtz-Dorten, 2017) at the time of admission and discharge of inpatient child and adolescent psychiatric treatment, and at 8, 24, and 37 weeks after discharge. Possible values range from 49 to 174 with higher scores indicating a worse outcome.
Change in symptom severity (parent report) | Admission, Pre (at discharge), Post (8 weeks after discharge), FollowUp1 (24 weeks after discharge), FollowUp2 (37 weeks after discharge)
  Symptom severity as assessed by parents is measured using the Diagnostic System for Mental Disorders according to ICD-10 and DSM-5 for Children and Adolescents - III Screening questionnaire (DISYPS-III SCREEN; Döpfner & Görtz-Dorten, 2017) at the time of admission and discharge of inpatient child and adolescent psychiatric treatment, and at 8, 24, and 37 weeks after discharge. Possible values range from 49 to 174 with higher scores indicating a worse outcome.
Change in symptom severity (teacher report) | Admission, Pre (at discharge), Post (8 weeks after discharge), FollowUp1 (24 weeks after discharge), FollowUp2 (37 weeks after discharge)
  Symptom severity as assessed by teachers is measured using the Diagnostic System for Mental Disorders according to ICD-10 and DSM-5 for Children and Adolescents - III Screening questionnaire (DISYPS-III SCREEN; Döpfner & Görtz-Dorten, 2017) at the time of admission and discharge of inpatient child and adolescent psychiatric treatment, and at 8, 24, and 37 weeks after discharge. Possible values range from 49 to 174 with higher scores indicating a worse outcome.
Change in Patients' Health-related quality of life | Admission, Pre (at discharge), Post (8 weeks after discharge), FollowUp1 (24 weeks after discharge), FollowUp2 (37 weeks after discharge)
  Health-related quality of life as assessed by patients is measured using the Health Related Quality of Life Questionnaire for Children and Young People and their Parents (KIDSCREEN-27; KIDSCREEN Group Europe, 2006) at the time of admission and discharge of inpatient child and adolescent psychiatric treatment, and at 8, 24, and 37 weeks after discharge. Possible values range from 27 to 135 with higher scores indicating a better outcome.
Change in Parents' Health-related quality of life | Admission, Pre (at discharge), Post (8 weeks after discharge), FollowUp1 (24 weeks after discharge), FollowUp2 (37 weeks after discharge)
  Health-related quality of life as assessed by parents is measured using the Health Related Quality of Life Questionnaire for Children and Young People and their Parents (KIDSCREEN-27; KIDSCREEN Group Europe, 2006) at the time of admission and discharge of inpatient child and adolescent psychiatric treatment, and at 8, 24, and 37 weeks after discharge. Possible values range from 27 to 135 with higher scores indicating a better outcome.
Patients' Satisfaction with treatment | Post (8 weeks after discharge)
  Satisfaction with treatment as assessed by patients is measured using questionnaire versions based on the Questionnaire for the assessment of treatment (FBB; Mattejat & Remschmidt, 1999) at 8 weeks after discharge. Possible values range from 0 to 76 with higher scores indicating a better outcome.
Parents' Satisfaction with treatment | Post (8 weeks after discharge)
  Satisfaction with treatment as assessed by parents is measured using questionnaire versions based on the Questionnaire for the assessment of treatment (FBB; Mattejat & Remschmidt, 1999) at 8 weeks after discharge. Possible values range from 0 to 84 with higher scores indicating a better outcome.
Therapists' Satisfaction with treatment | Post (8 weeks after discharge)
  Satisfaction with treatment as assessed by therapists is measured using questionnaire versions based on the Questionnaire for the assessment of treatment (FBB; Mattejat & Remschmidt, 1999) at 8 weeks after discharge. Possible values range from 0 to 72 with higher scores indicating a better outcome.
Teachers' Satisfaction with treatment | Post (8 weeks after discharge)
  Satisfaction with treatment as assessed by teachers is measured using questionnaire versions based on the Questionnaire for the assessment of treatment (FBB; Mattejat & Remschmidt, 1999) at 8 weeks after discharge. Possible values range from 0 to 56 with higher scores indicating a better outcome.
Difference and change in percentage of readmissions | Post (8 weeks after discharge), FollowUp1 (24 weeks after discharge), FollowUp2 (37 weeks after discharge)
  The percentage of readmissions is obtained by analyzing internal hospital controlling data. The change of these percentages over time is considered and compared across the study groups.

SECONDARY OUTCOMES:
Change in patients' Stress Vulnerability | Admission, Pre (at discharge), Post (8 weeks after discharge), FollowUp1 (24 weeks after discharge), FollowUp2 (37 weeks after discharge)
  Patients' stress vulnerability is measured with the appropriate sub-scale of the Questionnaire for the Survey of Stress and Stress Coping in Childhood and Adolescence - Revision (SSKJ 3-8R; Lohaus, Eschenbeck, Kohlmann, & Klein-Heßling, 2018), at the time of admission and discharge of inpatient child and adolescent psychiatric treatment, and at 8, 24, and 37 weeks after discharge. Possible values range from 7 to 28 with higher scores indicating a worse outcome.
Change in patients' Stress Coping Strategies | Admission, Pre (at discharge), Post (8 weeks after discharge), FollowUp1 (24 weeks after discharge), FollowUp2 (37 weeks after discharge)
  Patients' stress coping strategies are measured with the appropriate sub-scales of the Questionnaire for the Survey of Stress and Stress Coping in Childhood and Adolescence - Revision (SSKJ 3-8R; Lohaus, Eschenbeck, Kohlmann, & Klein-Heßling, 2018), at the time of admission and discharge of inpatient child and adolescent psychiatric treatment, and at 8, 24, and 37 weeks after discharge. Possible values range from 30 to 150 with higher scores indicating a better outcome.
Change in patients' school related self-efficacy | Admission, Pre (at discharge), Post (8 weeks after discharge), FollowUp1 (24 weeks after discharge), FollowUp2 (37 weeks after discharge)
  School related self-efficacy from the perspective of patients is measured based on the mean value of items from the WIRKSCHUL scales (Schulbezogene Selbstwirksamkeitserwartung [School-related self-efficacy]; Schwarzer & Jerusalem, 1999), at the time of admission and discharge from inpatient child and adolescent psychiatric treatment, and at 8, 24, and 37 weeks after discharge. Possible values range from 8 to 40 with higher scores indicating a better outcome.
Change in patients' social self-efficacy | Admission, Pre (at discharge), Post (8 weeks after discharge), FollowUp1 (24 weeks after discharge), FollowUp2 (37 weeks after discharge)
  Social self-efficacy from the perspective of patients is measured based on the mean value of items from the WIRKSOZ scales (Selbstwirksamkeitserwartung im Umgang mit sozialen Anforderungen [Self-efficacy in dealing with social demands]; Schwarzer & Jerusalem, 1999), at the time of admission and discharge from inpatient child and adolescent psychiatric treatment, and at 8, 24, and 37 weeks after discharge. Possible values range from 8 to 40 with higher scores indicating a better outcome.
Change in parents' social self-efficacy | Admission, Pre (at discharge), Post (8 weeks after discharge), FollowUp1 (24 weeks after discharge), FollowUp2 (37 weeks after discharge)
  Self-efficacy from the perspective of parents is measured based on the mean of adequately adapted items from the WIRKLEHR scale (Skala Lehrer-Selbstwirksamkeit [Teacher Self-Efficacy Scale]; Schwarzer & Jerusalem, 1999), at the time of admission and discharge and at 8, 24, and 37 weeks after discharge. Possible values range from 8 to 40 with higher scores indicating a better outcome.
Change in teachers' self-efficacy | Admission, Pre (at discharge), Post (8 weeks after discharge), FollowUp1 (24 weeks after discharge), FollowUp2 (37 weeks after discharge)
  Self-efficacy from the perspective of teachers is measured based on the mean value of adequately adapted items from the WIRKLEHR scale (Skala Lehrer-Selbstwirksamkeit [Teacher Self-Efficacy Scale]; Schwarzer & Jerusalem, 1999), at the time of admission and discharge and at 8, 24, and 37 weeks after discharge. Possible values range from 10 to 50 with higher scores indicating a better outcome.
Change in Occupational well-being of teachers | Pre (at discharge), Post (8 weeks after discharge), FollowUp1 (24 weeks after discharge), FollowUp2 (37 weeks after discharge)
  Teachers' occupational well-being is measured using the scales Emotional Exhaustion and Enthusiasm for Teaching (Kunter, Baumert, Leutner, Terhart, Seidel, Dicke, et al., 2016) at the time of discharge from inpatient child and adolescent psychiatric treatment and at 8, 24, and 37 weeks after discharge. Possible values range from 5 to 15 with higher scores indicating a better outcome.
Patients' satisfaction with technical components | Post (8 weeks after discharge)
  Patients' satisfaction with technical components is measured using thematically adapted items of the System Usability Scale (SUS; Brooke, 1996) at 8 weeks after discharge. Possible values range from 0 to 100 with higher scores indicating a better outcome.
Parents' satisfaction with technical components | Post (8 weeks after discharge)
  Parents' satisfaction with technical components is measured using thematically adapted items of the System Usability Scale (SUS; Brooke, 1996) at 8 weeks after discharge. Possible values range from 0 to 100 with higher scores indicating a better outcome.
Teachers' satisfaction with technical components | Post (8 weeks after discharge)
  Teachers' satisfaction with technical components is measured using thematically adapted items of the System Usability Scale (SUS; Brooke, 1996) at 8 weeks after discharge. Possible values range from 0 to 100 with higher scores indicating a better outcome.
Therapists' satisfaction with technical components | Post (8 weeks after discharge)
  Therapists' satisfaction with technical components is measured using thematically adapted items of the System Usability Scale (SUS; Brooke, 1996) at 8 weeks after discharge. Possible values range from 0 to 100 with higher scores indicating a better outcome.
Change in Parental stress | Admission, Pre (at discharge), Post (8 weeks after discharge), FollowUp1 (24 weeks after discharge), FollowUp2 (37 weeks after discharge)
  Parental stress is measured using the Eltern-Belastungs-Inventar (EBI; Tröster, 2010 [i.e., German version of the Parenting Stress Index; Abidin, 1997]), at the time of the child's admission and discharge from inpatient child and adolescent psychiatric treatment, and at 8, 24, and 37 weeks after discharge. Possible values range from 48 to 240 with higher scores indicating a worse outcome.
Parental strain | Admission
  Parental strain is measured with the Brief Symptom Checklist (BSCL; Franke, 2017) at the time of the child's admission for inpatient child and adolescent psychiatric treatment. Possible values range from 53 to 265 with higher scores indicating a worse outcome.
Change in Competence self-concept of teachers in dealing with students | Pre (at discharge), Post (8 weeks after discharge), FollowUp1 (24 weeks after discharge), FollowUp2 (37 weeks after discharge)
  Teachers' competence self-concept is measured using the identically named scale (Kunz Heim, Trachsler, Rindlisbacher, & Nido, 2007) at the time of admission and discharge of the student from inpatient child and adolescent psychiatric treatment, as well as at 8, 24, and 37 weeks after discharge. Possible values range from 5 to 20 with higher scores indicating a better outcome.
Change in teachers' professional competence in dealing with mentally ill students | Pre (at discharge), Post (8 weeks after discharge), FollowUp1 (24 weeks after discharge), FollowUp2 (37 weeks after discharge)
  Teachers' professional competence in dealing with mentally ill students is measured exploratively using the mean score of a self-developed scale, based on self-developed items and items from different studies in the field of Mental Health Literacy (Daniszewski, 2013; Hatcher, 2018; Reinke, Stormont, Herman, Puri, & Goel, 2011) and from teacher survey studies (Blömeke, Kaiser, & Lehmann, 2010; Kunter et al., 2016; Schwarzer & Jerusalem, 1999) at the time of the student's discharge from inpatient child and adolescent psychiatric treatment and 8, 24, and 37 weeks after discharge. Possible values of the total scale range from 24 to 120 with higher scores indicating a better outcome.
Patients' expectation of change | Pre (at discharge)
  Patients' expectation of change in relation to the aftercare is measured using the mean value of 4 thematically adapted items from the "Patient's expectation of change" of the Questionnaire for Measuring Common Factors in Psychotherapy (FERT; Vollmann, 2010). Possible values range from 0 to 16 with higher scores indicating a better outcome.
Parents' expectation of change | Pre (at discharge)
  Parents' expectation of change in relation to the aftercare is measured using the mean value of 4 thematically adapted items from the scale "Patient's expectation of change" of the Questionnaire for Measuring Common Factors in Psychotherapy (FERT; Vollmann, 2010). Possible values range from 0 to 16 with higher scores indicating a better outcome.

OTHER OUTCOMES:
Change in well-being (patients' Ambulatory Assessment) | Daily 2 weeks before discharge until 8 weeks after
  In the ambulatory assessment, children and adolescents provide information on their general well-being (pilot study). Possible values range from 1 to 5 with higher scores indicating a better outcome.
Change in affect (patients' Ambulatory Assessment) | Daily 2 weeks before discharge until 8 weeks after
  In the ambulatory assessment, children and adolescents provide information on their affect (Könen, Dirk, Leonhardt, & Schmiedek, 2016). Possible values range from 12 to 60 with higher scores indicating a better outcome.
Change in sleep quality (patients' Ambulatory Assessment) | Daily 2 weeks before discharge until 8 weeks after
  In the ambulatory assessment, children and adolescents provide information on their sleep quality (Könen et al., 2016). Possible values range from 2 to 10 with higher scores indicating a better outcome.
Change in percentage of school absenteeism (patients' Ambulatory Assessment) | Daily 2 weeks before discharge until 8 weeks after
  In the ambulatory assessment, children and adolescents provide information on their school absenteeism. Possible values range from 0 to 100 percent of absent days, with higher scores indicating a better outcome.
Change in school days (patients' Ambulatory Assessment) | Daily 2 weeks before discharge until 8 weeks after
  In the ambulatory assessment, children and adolescents provide information on their school days (KIDSCREEN Group Europe, 2006; Neubauer, Schmidt, Schmiedek, & Dirk, 2020). Possible values range from 4 to 20 with higher scores indicating a better outcome.
Change in relationship with peers (patients' Ambulatory Assessment) | Daily 2 weeks before discharge until 8 weeks after
  In the ambulatory assessment, children and adolescents provide information on their relationships with peers (Schmidt, Dirk, & Schmiedek, 2019). Possible values range from 4 to 20 with higher scores indicating a better outcome.
Change in relationship with parents (patients' Ambulatory Assessment) | Daily 2 weeks before discharge until 8 weeks after
  In the ambulatory assessment, children and adolescents provide information on their relationships with their parents (adapted from Schmidt, Dirk, & Schmiedek, 2019). Possible values range from 4 to 20 with higher scores indicating a better outcome.
Change in relationship with teachers (patients' Ambulatory Assessment) | Daily 2 weeks before discharge until 8 weeks after
  In the ambulatory assessment, children and adolescents provide information on their relationships with their teachers (adapted from KIDSCREEN Group Europe, 2006). Possible values range from 1 to 5 with higher scores indicating a better outcome.
Change in well-being (parents' Ambulatory Assessment) | Daily 2 weeks before discharge until 8 weeks after
  In the ambulatory assessment, parents provide data on their own general well-being (pilot study). Possible values range from 1 to 5 with higher scores indicating a better outcome.
Change in affect (parents' Ambulatory Assessment) | Daily 2 weeks before discharge until 8 weeks after
  In the ambulatory assessment, parents provide data on their affect (Könen et al., 2016). Possible values range from 12 to 60 with higher scores indicating a better outcome.
Change in child's well-being (parents' Ambulatory Assessment) | Daily 2 weeks before discharge until 8 weeks after
  In the ambulatory assessment, parents provide data on their child's well-being (pilot study). Possible values range from 1 to 5 with higher scores indicating a better outcome.
Change in relationship with the child (parents' Ambulatory Assessment) | Daily 2 weeks before discharge until 8 weeks after
  In the ambulatory assessment, parents provide data on their relationship with the child (adapted from Schmidt et al., 2019).Possible values range from 2 to 10 with higher scores indicating a better outcome.
Change in perceived support received from the clinic (teachers' Ambulatory Assessment) | Daily 2 weeks before discharge until 8 weeks after
  In the ambulatory assessment, teachers provide data on the perceived support they received from the clinic (self-development). Possible values range from 1 to 5 with higher scores indicating a better outcome.
Change in well-being (teachers' Ambulatory Assessment) | Daily 2 weeks before discharge until 8 weeks after
  In the ambulatory assessment, teachers provide data on their well-being (self-developed). Possible values range from 2 to 10 with higher scores indicating a better outcome.
Change in well-being of the student (teachers' Ambulatory Assessment) | Daily 2 weeks before discharge until 8 weeks after
  In the ambulatory assessment, teachers provide data on the well-being of the student (self-developed). Possible values range from 1 to 5 with higher scores indicating a better outcome.
Change in the teacher-student relationship (teachers' Ambulatory Assessment) | Daily 2 weeks before discharge until 8 weeks after
  In the ambulatory assessment, teachers provide data on the teacher-student relationship (adapted from KIDSCREEN Group Europe, 2006). Possible values range from 2 to 10 with higher scores indicating a better outcome.
Change in the school day (teachers' Ambulatory Assessment) | Daily 2 weeks before discharge until 8 weeks after
  In the ambulatory assessment, teachers provide data on the school day (KIDSCREEN Group Europe, 2006; Neubauer et al., 2020). Possible values range from 3 to 15 with higher scores indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias J. Renner, Prof. Dr., Study Director — University Hospital of Tuebingen, Germany; Caterina Gawrilow, Prof. Dr., Study Director — Department of Psychology, University of Tuebingen, Germany; Kelava Augustin, Prof. Dr., Study Director — Method Center, University of Tuebingen, Germany; Annette Conzelmann, Prof. Dr., Principal Investigator — University Hospital of Tuebingen, Germany; Dürrwächter Ute, Dr., Principal Investigator — University Hospital of Tuebingen, Germany; Schmid Johanna, Dr., Principal Investigator — University Hospital of Tuebingen, Germany; Kühnhausen Jan, Dr., Principal Investigator — University Hospital of Tuebingen, Germany; Finkbeiner Marlene, Principal Investigator — University Hospital of Tuebingen, Germany
Locations (1):
- Department of Child and Adolescent Psychiatry, Psychosomatics and Psychotherapy, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abidin RR. Parenting Stress Index: A measure of the parent-child system. Zalaquett CP, Wood RJ, editors. Lanham Maryland, USA: Scarecrow Education; 1997.
- [Background] Blömeke S, Kaiser G, Lehmann R. TEDS-M 2008. Professionelle Kompetenz und Lerngelegenheiten angehender Primarstufenlehrkräfte im internationalen Vergleich. Münster, Germany: Waxmann; 2010.
- [Background] Brooke J. SUS - a quick and dirty usability scale. In: Jordan PW, Thomas B, Weerdmeester, BA, McClelland IL, editors. Usability Evaluation in Industry. London, UK: Taylor & Francis; 1996. p. 189-94.
- [Background] Daniszewski TD. Teachers' mental health literacy and capacity towards student mental health. Electronic Thesis and Dissertation Repository. 2013:1165. https://ir.lib.uwo.ca/etd/1165
- [Background] Döpfner M, Görtz-Dorten A. Diagnostik-System für psychische Störungen nach ICD-10 und DSM-5 für Kinder und Jugendliche - III (DISYPS-III). Göttingen, Germany: Hogrefe; 2017.
- [Background] Franke GH. Brief-Symptom-Checklist (BSCL). Göttingen, Germany: Hogrefe; 2017.
- [Background] Hatcher AK. Measuring mental health literacy in education. Electronic Thesis and Dissertation Repository. 2018:5313. https://ir.lib.uwo.ca/etd/5313
- [Background] Konen T, Dirk J, Leonhardt A, Schmiedek F. The interplay between sleep behavior and affect in elementary school children's daily life. J Exp Child Psychol. 2016 Oct;150:1-15. doi: 10.1016/j.jecp.2016.04.003. Epub 2016 May 25. PMID 27236036
- [Background] Kunter M, Baumert J, Leutner D, Terhart E, Seidel T, Dicke T, et al. Dokumentation der Erhebungsinstrumente der Projektphasen des BilWiss-Forschungsprogramms von 2009 bis 2016. Frankfurt am Main, Germany: Goethe-Universität Frankfurt; 2016.
- [Background] Kunz Heim D, Trachsler E, Rindlisbacher S, Nido M. Schulen als Lernumgebungen für Lehrerinnen und Lehrer: Zusammenhänge zwischen Schulkontext, persönlichen Merkmalen und dem Weiterlernen von Lehrpersonen. Kreuzlingen, Switzerland: Pädagogische Hochschule Thurgau; 2007.
- [Background] Lohaus A, Eschenbeck H, Kohlmann C-W, Klein-Heßling J. Fragebogen zur Erhebung von Stress und Stressbewältigung im Kindes- und Jugendalter - Revision (SSKJ 3-8 R). Göttingen, Germany: Hogrefe; 2018.
- [Background] Mattejat F, Remschmidt H. Fragebogen zur Beurteilung der Behandlung (FBB). Göttingen, Germany: Hogrefe; 1999.
- [Background] Neubauer A, Schmidt A, Schmiedek F, Dirk J. Dynamic Reciprocal Relations of Achievement Goal Orientations with Daily Experiences of Success and Failure: An Ambulatory Assessment Study. 2020; doi:10.31234/osf.io/uypex.
- [Background] Reinke WM, Stormont M, Herman KC, Puri R, Goel N. Supporting children's mental health in schools: Teacher perceptions of needs, roles, and barriers. School Psychology Quarterly. 2011;26:1-13.
- [Background] Schmidt A, Dirk J, Schmiedek F. The importance of peer relatedness at school for affective well-being in children: Between-and within-person associations. Social Development. 2019;28:873-92.
- [Background] Schwarzer R, Jerusalem M. Skalen zur Erfassung von Lehrer- und Schülermerkmalen: Dokumentation der psychometrischen Verfahren im Rahmen der Wissenschaftlichen Begleitung des Modellversuchs Selbstwirksame Schulen. Berlin, Germany: Universität Berlin; 1999.
- [Background] The KIDSCREEN Group Europe. The KIDSCREEN-27 Questionnaire - Quality of life questionnaire for children and adolescents. Lengerich, Germany: Pabst Science Publishers; 2006.
- [Background] Tröster H. Eltern-Belastungs-Inventar (EBI): Deutsche Version des Parenting Stress Index (PSI) von R. R. Abidin. Göttingen, Germany: Hogrefe; 2010.
- [Background] Vollmann K. Construction and evaluation of a questionnaire for measuring common factors in psychotherapy (FERT) [dissertation]. Tuebingen, Germany: University Tuebingen; 2010 [Available from: http://nbn-resolving.de/urn:nbn:de:bsz:21-opus-47705].
- [Derived] Finkbeiner M, Kuhnhausen J, Schmid J, Conzelmann A, Durrwachter U, Wahl LM, Kelava A, Gawrilow C, Renner TJ. E-Mental-Health aftercare for children and adolescents after partial or full inpatient psychiatric hospitalization: study protocol of the randomized controlled DigiPuR trial. Trials. 2022 Aug 26;23(1):713. doi: 10.1186/s13063-022-06508-1. PMID 36028894